CLINICAL TRIAL: NCT01523288
Title: The Intestinal Function in People With Prader-Willi Syndrome
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Louise Kuhlmann Frandsen, Principal Investigator, Aarhus University Hospital
Other Study IDs: PWS-1051
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Prader-Willi Syndrome; Constipation; Incontinence
MeSH Terms: conditions — Prader-Willi Syndrome; Constipation

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prader-Willi patients
- Control group: Control group for ultrasound scan

SUMMARY:
The projects aim is to investigate the intestinal function of patients suffering from Prader-Willi Syndrome. The methods used are ultrasonographic measurement of the rectal diameter and gastrointestinal transit time

DETAILED DESCRIPTION:
Prader-Willi Syndrome (PWS) is a congenital genetical disease characterized by moderate retardation, food-seeking behavior and a serious risk of developing health threatening overweight, low stature, abnormal body composition and a lack of growth- and sex-hormones. They can not live an independent life and are reliant of help from care personnel.

People with PWS react abnormally to signals from their own bodies. E.g. they have a reduced sense of pain and can have a lacking urge to urination despite a full bladder. Most of the patients also have a relatively slow pulse, which can be consistent with a dysfunction in the nervous system (the parasympathetic nervous system) which also has large significance for the bladder- and bowel function.

The Intestinal function in people with PWS is a sparse described subject, which has not been systematically examined in scientific context. We therefore want to examine whether the bowel function in people with PWS are different from the bowel function in healthy people.

The subject is elucidated by a medical examination, a questionnaire, a registration of toilet habits, a measurement of the rectal diameter by an ultrasound scan and a measurement of the colonic transit time.

The results will be compared to findings in normal healthy people. Because no normal material exists for rectal diameter measured by ultrasound, we will establish one.

The result of the project will increase our knowledge of possible bowel dysfunctions such as constipation, in people with PWS and can immediately lead to improved care for and optimized treatment of the patients.

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* >14 days since last antibiotic treatment
* >14 days since last laxative treatment
* PWS confirmed genetically

Exclusion Criteria:

* previous abdominal surgery (except appendectomy or haemorrhoidectomy
* patient not capable of understanding the information
* treatment with eltroxin or antipsychotic medication
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Prader-Willi Syndrome
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Colonic Transit time | 6 days
  Measured ad modum Göteborg
Rectal diameter | 1 day
  measured by ultrasound scan

CONTACTS AND LOCATIONS:
Overall Officials: Louise K Frandsen, Stud.med, Principal Investigator — Centre of Rare Diseases, Pediatrics department, Aarhus University Hospital Skejby; Stense Farholt, Ph.D, Study Chair — Centre for Rare Diseases, Pediatrics department, Aarhus University Hospital Skejby; Klaus Krogh, DMSc, Study Chair — Medical Hepato-gastroenterological department, Aarhus University Hospital, Aarhus Sygehus; Iben M Jønsson, Ph.D, Study Chair — Pediatrics department, Aarhus University Hospital Skejby; Jens B Froekjaer, PhD, Study Chair — Department of Radiology, Aalborg Hospital
Locations (1):
- Centre of Rare Diseases, Pediatric department, Aarhus University Hospital Skejby, Aarhus, Aarhus N, Denmark